CLINICAL TRIAL: NCT04762498
Title: A Phase 4, Open-Label, Multicenter, Efficacy, Safety, Pharmacokinetics and Pharmacodynamics Trial of Intravenous KRYSTEXXA® (Pegloticase) Administered Every 4 Weeks With Co-Administration of Weekly Doses of Methotrexate in Patients With Uncontrolled Refractory Gout (FORWARD Open-Label [OL] Trial)
Brief Title: A Phase 4, Open-label Study of KRYSTEXXA® (Pegloticase) Co-administered With Methotrexate (MTX) in Patients With Uncontrolled Gout (FORWARD OL)
Acronym: FORWARD OL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-KRY-408
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Uncontrolled Gout; Chronic Gout
Keywords: Gout; KRYSTEXXA; Pegloticase; Methotrexate; Uncontrolled gout
MeSH Terms: conditions — Gout | interventions — Pegloticase; Methotrexate

STUDY DESIGN:
Intervention Model Description: Screening period up to 35 days, followed by 4-week methotrexate (MTX) tolerability run-in. Treatment consists of pegloticase IV Q4 Wks dose for a total of 6 infusions (24 Weeks) with co-administered weekly oral MTX. Optional extension treatment (24-48 weeks) will be available for 6 more infusions (total of 12). Study will consist of Cohort 1: 16 mg pegloticase, co-administered with weekly doses of oral MTX; and, potential Cohort 2: 24 to 32 mg pegloticase, co-administered with weekly doses of oral MTX and/or potential infusion duration reduction to 60 min.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegloticase 16mg cohort (Experimental): 16 mg IV dose of pegloticase q4 weeks with 15 mg methotrexate (MTX) weekly
  Interventions: Biological: Pegloticase; Drug: Methotrexate (MTX)
- Pegloticase 24/32mg cohort (Experimental): 24 to 32 mg IV dose of pegloticase q4 weeks with 15 mg MTX weekly
  Interventions: Biological: Pegloticase; Drug: Methotrexate (MTX)

INTERVENTIONS:
Biological: Pegloticase — IV dose of pegloticase q4 weeks co-administered with weekly oral methotrexate
Drug: Methotrexate (MTX) — 15 mg oral dose methotrexate administered weekly

SUMMARY:
This trial is to assess efficacy, safety, blood levels and bodily effects of up to 2 dose levels of intravenous (IV) pegloticase (KRYSTEXXA) infusions at every 4 week intervals (Q4 Weeks) for up to 6 months (Day 1 to 24 weeks with an optional 24 - 48 weeks treatment duration) when given in combination with weekly oral doses of methotrexate (MTX). The goal is to identify an appropriate dose to be administered every 4 weeks to be used for future clinical trials for patients with chronic gout that does not adequately respond to conventional therapy.

DETAILED DESCRIPTION:
The primary objective is to choose a dose for further investigation by assessing the effect of up to 2 dose levels of pegloticase administered IV Q4 weeks, co-administered with weekly doses of oral MTX, as measured by the sustained normalization of serum uric acid (sUA) to < 6 mg/dL for at least 80% of the time during Month 6 and the duration of sUA to < 6 mg/dL over 24 week treatment period in adult participants with chronic gout refractory to conventional therapy.

Acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent.
2. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.
3. Adult men or women ≥18 and <80 years of age.
4. Uncontrolled gout, defined as meeting the following criteria:

   * Hyperuricemia during the screening period defined as sUA ≥6 mg/dL, and;
   * Failure to maintain normalization of sUA with xanthine oxidase inhibitors at the maximum medically appropriate dose, or with a contraindication to xanthine oxidase inhibitor therapy based on medical record review or subject interview, and;
   * Symptoms of gout including at least 1 of the following:

     * Presence of at least one tophus
     * Recurrent flares defined as 2 or more flares in the past 12 months prior to screening
     * Presence of chronic gouty arthritis as evidenced by either clinical signs consistent with chronic synovitis on clinical examination or the presence of typical gouty erosion(s) on hand and/or foot X-rays
5. Willing to discontinue any oral urate lowering therapy for at least 7 days prior to MTX dosing at Week -4 and remain off while receiving pegloticase treatments.
6. Women of childbearing potential (including those with an onset of menopause <2 years prior to screening, non-therapy-induced amenorrhea for <12 months prior to screening, or not surgically sterile [absence of ovaries and/or uterus]) must have negative serum/urine pregnancy tests during Screening and Week -4; subjects must agree to use 2 reliable forms of contraception during the trial, one of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started ≥1 full cycle prior to Week -4 (start of MTX) and continue for 4 weeks/30 days after the last dose of pegloticase, or at least one ovulatory cycle after the last dose of MTX (whichever is the longest duration after the last dose of pegloticase or MTX). Highly effective contraceptive methods (with a failure rate <1% per year), when used consistently and correctly, include implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, or vasectomized partner.
7. Men who are not vasectomized must agree to use appropriate contraception so as to not impregnate a female partner of reproductive potential during the trial, beginning with the initiation of MTX at Week -4 and continuing and for at least 3 months after the last dose of MTX.
8. Able to tolerate MTX 15 mg orally for 4 weeks (Week -4 through Day 1) prior to enrollment.

Exclusion Criteria:

1. Weight >160 kg (352 pounds) at Screening.
2. Any serious acute bacterial infection, unless treated and completely resolved with antibiotics at least 2 weeks prior to the Day 1 Visit.
3. Severe chronic or recurrent bacterial infections, such as recurrent pneumonia or chronic bronchiectasis.
4. Current or chronic treatment with systemic immunosuppressive agents such as MTX, azathioprine, or mycophenolate mofetil; prednisone ≥10 mg/day or equivalent dose of other corticosteroid on a chronic basis (3 months or longer) would also meet exclusion criteria.
5. History of any transplant surgery requiring maintenance immunosuppressive therapy.
6. Known history of hepatitis B virus surface antigen positivity or hepatitis B DNA positivity.
7. Known history of hepatitis C virus RNA positivity, unless treated and viral load is negative.
8. Known history of Human Immunodeficiency Virus (HIV) positivity.
9. Glucose-6-phosphate dehydrogenase deficiency (tested at the Screening Visit centrally or locally).
10. Chronic renal impairment defined as estimated glomerular filtration rate (eGFR) <40 mL/min/1.73 m^2 or currently on dialysis.
11. Non-compensated congestive heart failure or hospitalization for congestive heart failure within 3 months of the Screening Visit, uncontrolled arrhythmia, treatment for acute coronary syndrome (myocardial infarction or unstable angina), or uncontrolled blood pressure (>160/100 mmHg) prior to enrollment at Day 1.
12. Pregnant, planning to become pregnant, breastfeeding, planning to impregnate female partner, or not on an effective form of birth control, as determined by the Investigator.
13. Prior treatment with pegloticase, another recombinant uricase (rasburicase), or concomitant therapy with a polyethylene glycol-conjugated drug.
14. Known allergy to pegylated products or history of anaphylactic reaction to a recombinant protein or porcine product.
15. Contraindication to MTX treatment or MTX treatment considered inappropriate.
16. Known intolerance to MTX.
17. Receipt of an investigational drug within 4 weeks or 5 half-lives, whichever is longer, prior to MTX administration at Week -4 or plans to take an investigational drug during the trial.
18. Liver transaminase levels (AST or ALT) > 1.25 X upper limit of normal (ULN) or albumin < the lower limit of normal (LLN) at the Screening Visit.
19. Chronic liver disease.
20. White blood cell count <4000/µl, hematocrit <32 percent, or platelet count <75,000/µl.
21. Currently receiving systemic or radiologic treatment for ongoing cancer, excluding non-melanoma skin cancer.
22. History of malignancy within 5 years other than non-melanoma skin cancer or in situ carcinoma of cervix.
23. Diagnosis of osteomyelitis.
24. Known history of hypoxanthine-guanine phosphoribosyl-transferase deficiency, such as Lesch-Nyhan and Kelley-Seegmiller syndrome.
25. Unsuitable candidate for the trial, based on the opinion of the Investigator (e.g., cognitive impairment), such that participation might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or complete the trial.
26. Alcohol use in excess of 3 alcoholic beverages per week.
27. A known intolerance to all protocol standard gout flare prophylaxis regimens (i.e., subject must be able to tolerate at least one: colchicine and/or non-steroidal anti-inflammatory drugs and/or low dose prednisone ≤10 mg/day).
28. Current pulmonary fibrosis, bronchiectasis or interstitial pneumonitis. If deemed necessary by the Investigator, a chest X-ray may be performed during Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of Serum Uric Acid (sUA) Responders (sUA < 6 mg/dL) During Month 6 | Month 6 (Weeks 20, 21, 22, 23, and 24)
  Responders are defined as participants achieving and maintaining sUA < 6 mg/dL for at least 80% of the time during Month 6. Participants meeting the sUA discontinuation criteria (pre-infusion sUA >6 mg/dL at 2 consecutive scheduled trial visits beginning with the Week 1 Visit) were counted as non-responders.
Time to first sUA ≥6 mg/dL after first achieving sUA <6 mg/dL, from the first pegloticase infusion until Week 24 | Day 1 to Week 24

SECONDARY OUTCOMES:
Pharmacokinetic parameters (e.g., AUC and, Cmax) | Baseline to Week 48
Proportion of subjects with pre-infusion sUA <6 mg/dL at each scheduled visit | Baseline to Week 48
Area under the sUA concentration vs time curve from Day 1 to Week 24 and Day 1 to Week 48 | Day 1 to Week 24 and Day 1 to Week 48
Proportion of the subjects sustained sUA< 6 mg/dL from Day 1 to Week 24 and Day 1 to Week 48 | Day 1 to Week 24 and Day 1 to Week 48
Proportion of subjects with anti-uricase antibodies and the proportion of subjects with anti-poly (ethylene glycol) antibodies and their titers at each scheduled visit | Baseline to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen; Supra Verma, MD, Study Director — Horizon Therapeutics
Locations (12):
- United States (12):
  - Orthopedic Physicians Alaska, Anchorage, Alaska
  - Arizona Arthritis & Rheumatology Research, PLLC, Glendale, Arizona
  - East Bay Rheumatology Medical Group, Inc., San Leandro, California
  - ProHealth Research Center, Doral, Florida
  - Napa Research Center, Pompano Beach, Florida
  - GCP Clinical Research, Tampa, Florida
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Shelby Clinical Research, LLC, Shelby, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Biopharma Informatic, LLC, Houston, Texas
  - Arthritis Clinic: Western Washington Medical Group, Bothell, Washington
  - Arthritis Northwest PLLC, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com